CLINICAL TRIAL: NCT01785927
Title: Clinical Trial Phase I of Antituberculosis Dry Powder Aerosols
Brief Title: The Safety of Tuberculosis Treatments by Oral Inhalation
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Principal Investigator, Teerapol Srichana, Associate Professor, Prince of Songkla University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RES.no. 18/2554
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Healthy
Keywords: Antituberculosis; Dry powder aerosols; Inhalation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- ABCD (Other): ABCD A = rifampicin, B = isoniazid, C= pyrazinamide, D = levofloxacin
  Interventions: Other: ABCD
- BCDA (Other): BCDA A = rifampicin, B = isoniazid, C= pyrazinamide, D = levofloxacin
  Interventions: Other: ABCD
- CDAB (Other): CDAB A = rifampicin, B = isoniazid, C= pyrazinamide, D = levofloxacin
  Interventions: Other: ABCD
- DABC (Other): DABC A = rifampicin, B = isoniazid, C= pyrazinamide, D = levofloxacin
  Interventions: Other: ABCD

INTERVENTIONS:
Other: ABCD — Rifampicin, isoniazid, pyrazinamide, and levofloxacin dry powders will be administered to each patient by randomization. Each formulation will be assigned the code, such as A, B, C, or D, and the treatment sequences will be generated as ABCD (sequence 1), BCDA (sequence 2), CDAB (sequence 3) and DABC (sequence 4). On the first day of drug dosing in period I, volunteers will be randomly assigned to a sequence of treatments as indicated in a pre-printed randomization scheme, which was generated using block randomization with block sizes of 4 and 6, and the allocation ratio of 1:1. Subjects will be stratified by sex. Subjects in sequence 1 will receive treatment A during the first study period and will then cross over to receive treatment B, C, and D at the second, third and fourth periods, respectively (each after a 7-day washout period).

SUMMARY:
The inhaled route of delivery has always been associated with the considerable challenge of getting the drug to its target. The lungs are a highly complex organ designed to filter inspired air, with many different cell types contributing to their function. Furthermore, the lungs may change dramatically when afflicted by disease resulting in an internal environment that works against the drug reaching and interacting successfully with the target. For targets in the upper airways this will have lesser significance, but drug delivery to the deep lung may be impeded by changes such as mucus hyper-secretion or thickening or airway narrowing.

In order to interpret toxicology findings it is necessary to reconcile test sensitivity, background biological variation, normal responses to inhaled materials and drug or medicine-specific adverse effects. Identification of adverse end-points is an area where better control data sets might help discern true adverse effects from a normal physiological lung response. The lung responds acutely to inhalation of irritant materials by hyper-secretion of mucus, chemokine release, inflammatory cell recruitment and cough and collectively these may be characterized as non-specific irritancy.

DETAILED DESCRIPTION:
Four formulations of antituberculosis drug (rifampicin, isoniazid, pyrazinamide, and levofloxacin) will be administered to each patient by randomization. Each formulation will be assigned the code, such as A, B, C, or D, and the treatment sequences will be generated as ABCD (sequence 1), BCDA (sequence 2), CDAB (sequence 3) and DABC (sequence 4). On the first day of drug dosing in period I, volunteers will be randomly assigned to a sequence of treatments as indicated in a pre-printed randomization scheme, which was generated using block randomization with block sizes of 4 and 6, and the allocation ratio of 1:1. Subjects will be stratified by sex. Subjects in sequence 1 will receive treatment A during the first study period and will then cross over to receive treatment B, C, and D at the second, third and fourth periods, respectively (each after a 7-day washout period).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45 years
* Body mass index 18-27 kg/m2
* Healthy
* In the case of reproductive age woman, effective contraceptive will be used for at least 4 weeks prior to a screening examination until the end of study.
* Non-lactating women
* Patients who are willing to participate in the trial and will first sign the informed consent form.

Exclusion Criteria:

* Allergic to any antituberculosis drugs or other components
* High blood pressure (diastolic pressure > 90 mmHg)
* Liver enzymes (AST and ALT) > 2 times of upper normal value
* Pregnancy or lactation
* No underlying diseases such as asthma, COPD, chronic kidney disease, diabetes mellitus, liver disease, immunocompromised deficiency, etc.
* HBsAg positive
* Abnormality in chest X-ray or routine laboratory tests
* Smokers > 10 cigarette/day or smokers < 10 cigarettes/day who could not quit at least 7 days before study and throughout study (including the washout between periods)
* Regular alcohol consumption (more than 1 time/week) or alcohol consumption within 7 days prior to the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Cytokine levels (Tumor Necrosis Factor-α and Interleukin-1β) | Two months

SECONDARY OUTCOMES:
Liver function tests (tB/dB, AST, ALT, ALP) | Two months

OTHER OUTCOMES:
Adverse events | Two months

CONTACTS AND LOCATIONS:
Locations (1):
- Songklanagarind Hospital, Hat Yai, Changwat Songkhla, Thailand